CLINICAL TRIAL: NCT04944420
Title: Evaluating an App-based Treatment for Distressed Caregivers of Persons With Moderate Dementia: Health enSuite Caregivers Study
Brief Title: Health enSuite Caregivers: an App-based Treatment for Distressed Caregivers of Persons With Moderate Dementia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Patrick J. McGrath, Principal Investigator, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1026747
Record Dates: First submitted 2021-06-14; First posted 2021-06-29 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-08

CONDITIONS: Caregiver Burnout
Keywords: Caregiver Burnout; Caregiver Stress; Caregivers; Dementia
MeSH Terms: conditions — Caregiver Burden; Dementia

STUDY DESIGN:
Intervention Model Description: This project consists of a pragmatic randomized controlled trial (RCT). The Consolidated Standards of Reporting Trials (CONSORT) recommendations (http://www.consort-statement.org/) will be used to guide the methodology. Participants will be randomly allocated in a 1:1 ratio to either the intervention group or a waitlist control group. Participants in both groups will complete self-assessments, including key outcome measures, at baseline, and 2-, and 5-months post-randomization. Participants in the intervention group will receive the full Health enSuite Caregivers program described below immediately after being randomized to this group.
  Participants in the control group will be waitlisted and receive only treatment as usual during the study. After their participation is the study has ended, participants in the control group will be given access to the full Health enSuite Caregivers program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention group will have access to Health enSuite Caregivers, an e-health program designed to meet some of the most common needs of caregivers of persons with dementia, including information about dementia and dementia care, caregivers' emotional health, formal or informal help received from others. It also recommends specific strategies to promote well-being and provides tools to help caregivers implement these strategies in their everyday lives.
  Health enSuite Caregivers is designed to offer advice to caregivers of persons with dementia based on an assessment of their specific needs. Topics are divided into five main content areas, which are recommended based on an assessment of the caregivers current challenges and sources of stress.
  Interventions: Behavioral: Health enSuite Caregivers
- Waitlist Control (No Intervention): Participants in the control group will be waitlisted and receive only treatment as usual during the study. After their participation is the study has ended, participants in the control group will be given access to the full Health enSuite Caregivers program.

INTERVENTIONS:
Behavioral: Health enSuite Caregivers — Advice within Health enSuite Caregivers is organized into 5 priority areas: Taking Care of Yourself (Self-care), Support for You (Support), Supporting the Person Living with Dementia (Characteristics of Persons Living with Dementia), Communication, and Time Management.
  Under "My Priority Areas", participants will see these in order from highest to lowest need, based on their answers to the needs assessment. Each priority area contains small subtopics and specific tips for things to "Try" or "Avoid". Navigation through the priority areas is user directed and at the participant's discretion. The goal is to make the information they need easy to access.
  Arms: Intervention

SUMMARY:
Health enSuite Caregivers is an e-health program designed to meet some of the most common needs of caregivers of persons with dementia, including information about dementia and dementia care, caregivers' emotional health, formal or informal help received from others. It also recommends specific strategies to promote wellbeing and provides tools to help caregivers implement these strategies in their everyday lives. Health enSuite Caregivers is available online and as a smartphone app. Its development was informed by reviews of caregivers' needs and existing commercially available apps F. A systematic search of commercially available smartphone applications for caregivers found that many apps did not consider each caregiver's unique needs and were limited to psychoeducational content (no tools for self-management). Furthermore, most existing programs have not been rigorously tested or lack evidence to support their effectiveness.

DETAILED DESCRIPTION:
As the Canadian population ages, the demand for informal caregivers is expected to increase. Currently, an estimated 8 million Canadians provide unpaid assistance and ongoing care to family members and friends in need of support due to physical, cognitive, or mental health conditions. Challenges associated with being an informal caregiver vary based on a number of factors including how much time is involved, the health of the person being cared for, and the care needs. Although all caregivers may experience distress, caregivers of people with dementia are at especially high risk for psychological distress and poor health outcomes. Nearly half of the individuals who are providing care for someone with dementia experience symptoms of distress.

It is important to provide caregivers with information and support so that they can manage these demands without compromising their own wellbeing. However, existing programs for caregivers are relatively limited. Primary care providers play an important role in supporting caregivers of people with dementia; however, there is a lack of effective, easily accessible programs for primary healthcare providers to recommend to a distressed caregiver of someone with dementia. We developed Health enSuite Caregivers as a potential solution to this problem.

ELIGIBILITY:
To be eligible for this trial, participants will have to satisfy the following criteria:

1. The participant is 18 years or older.
2. The participant has regular access to an internet connected device (e.g., smartphone, tablet, or computer).
3. The participant is a caregiver of a person with moderate dementia.
4. The participant provides a least one hour of care per week.
5. The participant is experiencing distress associated with caregiving (score DQ5 >= 11).

Rational:

Health enSuite Caregivers program being tested in this trial requires the use of an internet connected device. Health enSuite Caregivers can be downloaded as a mobile application for use on a smartphone or tablet, or it can be accessed through the web browser on an electronic device with an internet connection. People who do not have regular access to an internet connected device are unlikely to benefit from Health enSuite Caregivers, and therefore they will be excluded.

Health enSuite Caregivers is designed to help primary caregivers of persons with moderate dementia. Therefore, the eligibility screening questionnaire includes items to assess dementia severity. To ensure that the participants has ongoing caregiving duties, they must self-report providing at least one hour of care per week. There is no clear consensus on the number of hours of care that all primary caregivers provide. Reports from the Canadian Institute for Health Informatics estimate that on average informal caregivers of persons with dementia provide 26 hours of care per week (3). One hour per week was selected as a minimum threshold to exclude people with very limited caregiving responsibilities.

Health enSuite Caregivers is intended to help caregivers who are experiencing some degree of distress. Participants must also score above the cut-off score (>=11) for distress on the DQ-5 (18), a population distress screening measure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Carer wellbeing | Baseline assessment, 2 months post randomization, 5 months post randomization
  Carer wellbeing in terms of emotional health and interpersonal relationships will be assessed as the primary outcome measure in this study using the Carer Wellbeing and Support Scales (CWS(9). It is recommended as the most appropriate instrument for the assessment of quality of life in informal carers of people with dementia (10). The CWS evaluates the multiple facets of well-being of people caring for someone with dementia. The aggregate of the responses to the questions under "your role as a carer", "your relationship with the person you care for", "your relationship with family and friends" and "your emotional well-being" will be used as the primary outcome in this RCT as these are the forms of wellbeing Health enSuite Caregivers is hypothesized to effect most strongly.

SECONDARY OUTCOMES:
Overall carer wellbeing and specific facets of carer welling | Baseline assessment, 2 months post randomization, 5 months post randomization
  Responses on the CWS will be used to compute several secondary outcomes that may be affected by Health enSuite Caregivers.
  * Total carer wellbeing (sum of all 33 items)
  * Your role as a carer (items 1-5)
  * Relationship with the PWD (items 6-11)
  * Relationships with friends and family (items 12-15)
  * Emotional wellbeing (items 21-26)
  * Financial wellbeing (items 16-18)
  * Physical health (items 19-20)
  * Stigma and discrimination (item 27)
  * Personal safety (item 28-29)
  * Safety of PWD (items 30-32)
Self-efficacy | Baseline assessment, 2 months post randomization, 5 months post randomization
  Caregiver self-efficacy will be measured using the family caregivers' self-efficacy for managing dementia scale (11). It measures the degree of confidence caregivers have about their ability to complete necessary caregiving tasks. It includes 10 items and is scored based on a 10-point Likert scale from 1 ("not at all certain") to 10 ("very certain"). This scale has been widely used in studies of caregivers of people with dementia and has been found to have good internal consistency (11-13).
Psychological distress | Baseline assessment, 2 months post randomization, 5 months post randomization
  The Distress Questionnaire-5 (DQ-5) (18) will be used to assess psychological distress among caregivers. This 5-item measure captures general emotional distress and has demonstrated strong psychometric properties. We hypothesize that participants assigned to the intervention group will report lower levels of psychological distress at both 2- and 5-months post-randomization compared to participants in the control group. Specifically, DQ-5 scores are expected to decrease from baseline to follow-up in the intervention group, reflecting a reduction in emotional distress over time.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick McGrath, Principal Investigator — IWK Health Centre

IPD SHARING:
Plan to Share IPD: Yes
De-identified data sets may be retained and stored within the Centre for Research in Family Health as required for future research or program development, if merited. During Consent, participants will be offered the option of allowing their de-identified study data to be re-used by other approved researchers under the conditions that the research projects are approved by an appropriate ethics board and the researchers sign an agreement ensuring confidentiality and restricting data use only to the approved study. A database will be created containing only the data for those participants who agree will be available to researchers who meet these criteria.
Time Frame: From study closure to five years post publication.
Access Criteria: During Consent, participants will be offered the option of allowing their de-identified study data to be re-used by other approved researchers under the conditions that the research projects are approved by an appropriate ethics board and the researchers sign an agreement ensuring confidentiality and restricting data use only to the approved study.

REFERENCES:
- [Background] Hango D. Insights on Canadian Society Support received by caregivers in Canada. Stat Canada. 2020;(75).
- [Background] Brodaty H, Donkin M. Family caregivers of people with dementia. Dialogues Clin Neurosci. 2009;11(2):217-28. doi: 10.31887/DCNS.2009.11.2/hbrodaty. PMID 19585957
- [Background] Canadian Institute for Health Information. Unpaid caregiver challenges and supports. 2018.
- [Background] Stall N. We should care more about caregivers. CMAJ. 2019 Mar 4;191(9):E245-E246. doi: 10.1503/cmaj.190204. No abstract available. PMID 30833490
- [Background] Queluz FNFR, Kervin E, Wozney L, Fancey P, McGrath PJ, Keefe J. Understanding the needs of caregivers of persons with dementia: a scoping review. Int Psychogeriatr. 2020 Jan;32(1):35-52. doi: 10.1017/S1041610219000243. PMID 30967164
- [Background] Wozney L, Freitas de Souza LM, Kervin E, Queluz F, McGrath PJ, Keefe J. Commercially Available Mobile Apps for Caregivers of People With Alzheimer Disease or Other Related Dementias: Systematic Search. JMIR Aging. 2018 Dec 7;1(2):e12274. doi: 10.2196/12274. PMID 31518255
- [Background] Duggleby W, Ploeg J, McAiney C, Peacock S, Fisher K, Ghosh S, Markle-Reid M, Swindle J, Williams A, Triscott JA, Forbes D, Jovel Ruiz K. Web-Based Intervention for Family Carers of Persons with Dementia and Multiple Chronic Conditions (My Tools 4 Care): Pragmatic Randomized Controlled Trial. J Med Internet Res. 2018 Jun 29;20(6):e10484. doi: 10.2196/10484. PMID 29959111
- [Background] Quirk A, Smith S, Hamilton S, Lamping D, Lelliott P, Stahl D, et al. Development of the carer well-being and support (CWS) questionnaire. Ment Heal Rev J. 2012 Sep 21;17(3):128-38.
- [Background] Dow J, Robinson J, Robalino S, Finch T, McColl E, Robinson L. How best to assess quality of life in informal carers of people with dementia; A systematic review of existing outcome measures. PLoS One. 2018 Mar 14;13(3):e0193398. doi: 10.1371/journal.pone.0193398. eCollection 2018. PMID 29538433
- [Background] Fortinsky RH, Kercher K, Burant CJ. Measurement and correlates of family caregiver self-efficacy for managing dementia. Aging Ment Health. 2002 May;6(2):153-60. doi: 10.1080/13607860220126763. PMID 12028884
- [Background] Gallagher D, Ni Mhaolain A, Crosby L, Ryan D, Lacey L, Coen RF, Walsh C, Coakley D, Walsh JB, Cunningham C, Lawlor BA. Self-efficacy for managing dementia may protect against burden and depression in Alzheimer's caregivers. Aging Ment Health. 2011 Aug;15(6):663-70. doi: 10.1080/13607863.2011.562179. Epub 2011 May 24. PMID 21547745
- [Background] Spitznagel MB, Tremont G, Davis JD, Foster SM. Psychosocial predictors of dementia caregiver desire to institutionalize: caregiver, care recipient, and family relationship factors. J Geriatr Psychiatry Neurol. 2006 Mar;19(1):16-20. doi: 10.1177/0891988705284713. PMID 16449755
- [Background] Keefe J, Guberman N, Fancey P, Barylak L, Nahmiash D. Caregivers' Aspirations, Realities, and Expectations: The CARE Tool. J Appl Gerontol. 2008 Jun 11;27(3):286-308.
- [Background] Michie S, Richardson M, Johnston M, Abraham C, Francis J, Hardeman W, Eccles MP, Cane J, Wood CE. The behavior change technique taxonomy (v1) of 93 hierarchically clustered techniques: building an international consensus for the reporting of behavior change interventions. Ann Behav Med. 2013 Aug;46(1):81-95. doi: 10.1007/s12160-013-9486-6. PMID 23512568
- [Background] Cheng ST, Li KK, Losada A, Zhang F, Au A, Thompson LW, Gallagher-Thompson D. The effectiveness of nonpharmacological interventions for informal dementia caregivers: An updated systematic review and meta-analysis. Psychol Aging. 2020 Feb;35(1):55-77. doi: 10.1037/pag0000401. PMID 31985249
- [Background] Qiu D, Hu M, Yu Y, Tang B, Xiao S. Acceptability of psychosocial interventions for dementia caregivers: a systematic review. BMC Psychiatry. 2019 Jan 14;19(1):23. doi: 10.1186/s12888-018-1976-4. PMID 30642300
- [Background] Batterham PJ, Werner-Seidler A, O'Dea B, Calear AL, Maston K, Mackinnon A, Christensen H. Psychometric properties of the Distress Questionnaire-5 (DQ5) for measuring psychological distress in adolescents. J Psychiatr Res. 2024 Jan;169:58-63. doi: 10.1016/j.jpsychires.2023.11.004. Epub 2023 Nov 18. PMID 38000185